CLINICAL TRIAL: NCT03375047
Title: A Phase 1/2, Randomized, Double-Blinded, Placebo-Controlled, Combined Single and Multiple Ascending Dose Study Evaluating the Safety, Tolerability, and Biological Activity of MRT5005 Administered by Nebulization to Adult Subjects With Cystic Fibrosis
Brief Title: Study to Evaluate the Safety & Tolerability of MRT5005 Administered by Nebulization in Adults With Cystic Fibrosis
Acronym: RESTORE-CF
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MRT5005-101
Record Dates: First submitted 2017-09-07; First posted 2017-12-15 (Actual); Results first posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; CF
MeSH Terms: conditions — Cystic Fibrosis | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Part A - SAD Group 1: MRT5005 8 mg (Experimental): Participants received single dose of MRT5005 8 milligrams (mg) by nebulization on Day 1.
  Interventions: Drug: MRT5005
- Part A - SAD Group 2: MRT5005 16 mg (Experimental): Participants received single dose of MRT5005 16 mg by nebulization on Day 1.
  Interventions: Drug: MRT5005
- Part A - SAD Group 3: MRT5005 20 mg (Experimental): Participants received single dose of MRT5005 20 mg by nebulization on Day 1.
  Interventions: Drug: MRT5005
- Part A - SAD Group 4: MRT5005 24 mg (Experimental): Participants received single dose of MRT5005 24 mg by nebulization on Day 1.
  Interventions: Drug: MRT5005
- Part A - SAD Groups: Pooled Placebo (Placebo Comparator): Participants received single dose of placebo (normal saline) by nebulization on Day 1. Data were analyzed as a pooled population for all participants who received placebo in Part A SAD groups and reported in this arm.
  Interventions: Drug: Normal saline
- Part B - MAD Group 1: MRT5005 8 mg (Experimental): Participants received MRT5005 8 mg once weekly by nebulization for 5 weeks (i.e., on Day 1, Day 8, Day 15, Day 22 and Day 29).
  Interventions: Drug: MRT5005
- Part B - MAD Group 2: MRT5005 12 mg (Experimental): Participants received MRT5005 12 mg once weekly by nebulization for 5 weeks (i.e., on Day 1, Day 8, Day 15, Day 22 and Day 29).
  Interventions: Drug: MRT5005
- Part B - MAD Group 3: MRT5005 16 mg (Experimental): Participants received MRT5005 16 mg once weekly by nebulization for 5 weeks (i.e., on Day 1, Day 8, Day 15, Day 22 and Day 29).
  Interventions: Drug: MRT5005
- Part B - MAD Group 4: MRT5005 20 mg (Experimental): Participants received MRT5005 20 mg once weekly by nebulization for 5 weeks (i.e., on Day 1, Day 8, Day 15, Day 22 and Day 29).
  Interventions: Drug: MRT5005
- Part B - MAD Groups: Pooled Placebo (Placebo Comparator): Participants received placebo (normal saline) once weekly by nebulization for 5 weeks (i.e., on Day 1, Day 8, Day 15, Day 22 and Day 29). Data were analyzed as a pooled population for all participants who received placebo in Part B MAD groups and reported in this arm.
  Interventions: Drug: Normal saline
- Part D: MRT5005 4 mg (Experimental): Participants received MRT5005 4 mg once daily by nebulization from Day 1 to Day 5.
  Interventions: Drug: MRT5005
- Part D: Placebo (Placebo Comparator): Participants received placebo (normal saline) once daily by nebulization from Day 1 to Day 5.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: MRT5005 — Nebulization of MRT5005
  Arms: Part A - SAD Group 1: MRT5005 8 mg; Part A - SAD Group 2: MRT5005 16 mg; Part A - SAD Group 3: MRT5005 20 mg; Part A - SAD Group 4: MRT5005 24 mg; Part B - MAD Group 1: MRT5005 8 mg; Part B - MAD Group 2: MRT5005 12 mg; Part B - MAD Group 3: MRT5005 16 mg; Part B - MAD Group 4: MRT5005 20 mg; Part D: MRT5005 4 mg
Drug: Normal saline — Normal Saline for Inhalation
  Arms: Part A - SAD Groups: Pooled Placebo; Part B - MAD Groups: Pooled Placebo; Part D: Placebo

SUMMARY:
This Phase 1/2, first-in-human study evaluated the safety and tolerability of single and multiple escalating doses of MRT5005 administered by nebulization to the respiratory tract of adult subjects with cystic fibrosis (CF).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CF as defined by both of the following:

  * Two CF disease-causing cystic fibrosis transmembrane conductance regulator (CFTR) mutations in Class I or II (genotype confirmed at the screening visit).
  * Chronic sinopulmonary disease and/or gastrointestinal/nutritional abnormalities consistent with CF disease.
* Clinically stable CF disease, as judged by the investigator.
* Forced expiratory volume in 1 second (FEV1) ≥50% and ≤90% of the predicted normal for age, gender, and height at screening.
* Resting oxygen saturation ≥92% on room air (pulse oximetry).

Exclusion Criteria:

* An acute upper or lower respiratory infection, pulmonary exacerbation, or clinically significant episode of hemoptysis or change in chronic respiratory medications (including antibiotics) for CF lung disease within 28 days prior to dosing with investigational product on Day 1.
* Participants were receiving treatment with ivacaftor monotherapy (KALYDECO).
* Parts A and B only: Were receiving treatment with triple combination therapy (TRIKAFTA).
* Participants with a Class III, IV, or V CFTR gene mutation in at least 1 allele.
* Infection with highly virulent bacteria associated with accelerated decline in pulmonary function and/or decreased survival (e.g., Burkholderia cenocepacia, Burkholderia dolosa, Mycobacterium abscessus).

Treatment with ORKAMBI or SYMDEKO was not an exclusion for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - National Jewish Health, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - Northwestern University, Chicago, Illinois
  - University of Indiana, Indianapolis, Indiana
  - Maine Medical Center, Portland, Maine
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health and Sciences University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - New Orleans Center for Clinical Research, Knoxville, Tennessee
  - University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Miah KM, Hyde SC, Gill DR. Emerging gene therapies for cystic fibrosis. Expert Rev Respir Med. 2019 Aug;13(8):709-725. doi: 10.1080/17476348.2019.1634547. Epub 2019 Jun 27. PMID 31215818

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 16 active centers. A total of 53 participants were screened from 10 May 2018 to 22 February 2021, of which 11 were screen failures. Screen failures were mainly due to not meeting the eligibility criteria.
Pre-assignment Details: Study consisted of 4 parts: Part A-single ascending dose (SAD), Part B-multiple ascending dose (MAD), Part C (bronchoscopy groups) and Part D (daily dosing). A total of 42 participants were randomized (3:1 ratio) in Parts A, B and D to receive either MRT5005 or placebo. Part C was removed from protocol in 3rd amendment (dated 29 July 2019) prior to any participant enrollment in Part C. Participants were allowed to take part in 1 part of study only and results of Parts A, B and D were reported.
Period: Overall Study
Arm/Group | Part A - SAD Group 1: MRT5005 8 mg | Part A - SAD Group 2: MRT5005 16 mg | Part A - SAD Group 3: MRT5005 20 mg | Part A - SAD Group 4: MRT5005 24 mg | Part A - SAD Groups: Pooled Placebo | Part B - MAD Group 1: MRT5005 8 mg | Part B - MAD Group 2: MRT5005 12 mg | Part B - MAD Group 3: MRT5005 16 mg | Part B - MAD Group 4: MRT5005 20 mg | Part B - MAD Groups: Pooled Placebo | Part D: MRT5005 4 mg | Part D: Placebo
Started | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 4 | 3 | 5 | 6 | 2
Completed | 3 | 3 | 2 | 3 | 4 | 3 | 3 | 3 | 3 | 4 | 6 | 2
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Site closure due to Coronavirus disease 2019 pandemic | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety analysis set included all randomized participants who received study treatment.
Groups:
- Part A - SAD Group 1: MRT5005 8 mg: Participants received single dose of MRT5005 8 mg by nebulization on Day 1.
- Total: Total of all reporting groups
Arm/Group | Part A - SAD Group 1: MRT5005 8 mg | Part A - SAD Group 2: MRT5005 16 mg | Part A - SAD Group 3: MRT5005 20 mg | Part A - SAD Group 4: MRT5005 24 mg | Part A - SAD Groups: Pooled Placebo | Part B - MAD Group 1: MRT5005 8 mg | Part B - MAD Group 2: MRT5005 12 mg | Part B - MAD Group 3: MRT5005 16 mg | Part B - MAD Group 4: MRT5005 20 mg | Part B - MAD Groups: Pooled Placebo | Part D: MRT5005 4 mg | Part D: Placebo | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 4 | 3 | 5 | 6 | 2 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 4 | 3 | 4 | 6 | 2 | 41
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 2 | 1 | 2 | 3 | 1 | 3 | 1 | 3 | 5 | 1 | 23
  Male | 3 | 2 | 1 | 2 | 2 | 0 | 2 | 1 | 2 | 2 | 1 | 1 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 3 | 5 | 6 | 2 | 41
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Parts A, B and D: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that did not necessarily had a causal relationship with the study treatment. A serious adverse event (SAE) was any untoward medical occurrence (whether considered to be related to study treatment or not) that at any dose: resulted in death; or was life-threatening; or required inpatient hospitalization or prolongation of existing hospitalization; or resulted in persistent or significant disability/incapacity; or was a congenital abnormality/birth defect; or was an important medical event. The TEAEs were defined as events that were newly reported or reported to worsen in severity after the start of study treatment up to 48 weeks (end of follow-up period) after the last dose of study treatment administration.
Time Frame: From the first dose of study treatment administration (Day 1) up to 48 weeks (end of the follow-up period) after the last dose of study treatment administration (Part A: Day 337, Part B: Day 365 and Part D: Day 341)
Population: The Safety analysis set included all randomized participants who received study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A - SAD Group 1: MRT5005 8 mg | Part A - SAD Group 2: MRT5005 16 mg | Part A - SAD Group 3: MRT5005 20 mg | Part A - SAD Group 4: MRT5005 24 mg | Part A - SAD Groups: Pooled Placebo | Part B - MAD Group 1: MRT5005 8 mg | Part B - MAD Group 2: MRT5005 12 mg | Part B - MAD Group 3: MRT5005 16 mg | Part B - MAD Group 4: MRT5005 20 mg | Part B - MAD Groups: Pooled Placebo | Part D: MRT5005 4 mg | Part D: Placebo
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 4 | 3 | 5 | 6 | 2
Participants
  Any TEAE | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 4 | 3 | 5 | 6 | 2
  Any Serious TEAE | 0 | 0 | 1 | 1 | 3 | 1 | 1 | 0 | 2 | 2 | 1 | 1

2. Secondary Outcome: Parts A, B and D: Absolute Change From Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1)
Description: Spirometry was performed according to the guidelines published by the American Thoracic Society for standardization of spirometry. The ppFEV1 was assessed during the spirometry testing. For Parts A and B, the baseline value was defined as the average of the results from testing on Day -1 and at pre-dose on Day 1. For Part D, the baseline value was defined as the result from testing pre-dose on Day 1. Here, Baseline= BL, Day= D, pre-dose= PrD, hours post dose= hPD.
Time Frame: Part A:BL, D1(8hPD), D2(24hPD), D3, D8, D15 and D29; Part B:BL, D1(6hPD), D2, D8(PrD and 6hPD), D9, D15(PrD and 6hPD), D16, D22(PrD and 6hPD), D23, D29(PrD and 6hPD), D30, D36, D43 and D57; Part D:BL, D1(2hPD), PrD on D2, D3, D4 and D5, D11, D18 and D32
Population: The Safety analysis set included all randomized participants who received study treatment. Only those participants with data collected at specified timepoints are reported. '0' in the number analyzed field denotes that the specific time point category is not applicable to the respective reporting arm.
Measure: Mean (Standard Deviation); unit: percent predicted FEV1
Arm/Group | Part A - SAD Group 1: MRT5005 8 mg | Part A - SAD Group 2: MRT5005 16 mg | Part A - SAD Group 3: MRT5005 20 mg | Part A - SAD Group 4: MRT5005 24 mg | Part A - SAD Groups: Pooled Placebo | Part B - MAD Group 1: MRT5005 8 mg | Part B - MAD Group 2: MRT5005 12 mg | Part B - MAD Group 3: MRT5005 16 mg | Part B - MAD Group 4: MRT5005 20 mg | Part B - MAD Groups: Pooled Placebo | Part D: MRT5005 4 mg | Part D: Placebo
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 4 | 3 | 5 | 6 | 2
percent predicted FEV1
  Day 1: 2 hours post-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2
  Day 1: 2 hours post-dose |  |  |  |  |  |  |  |  |  |  | 5.1117 (3.75481) | -2.4150 (1.23744)
  Day 1: 6 hours post-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 4 | 3 | 5 | 0 | 0
  Day 1: 6 hours post-dose |  |  |  |  |  | -2.7017 (3.37188) | -0.3417 (2.17959) | -0.0062 (2.66067) | -1.9533 (8.52538) | 1.8400 (4.62365) |  |
  Day 1: 8 hours post-dose: number analyzed (Participants) | 3 | 3 | 3 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 1: 8 hours post-dose | 3.6550 (0.94230) | 7.2233 (7.29017) | 1.1067 (1.91247) | 2.4525 (0.44194) | 1.1088 (3.58541) |  |  |  |  |  |  |
  Day 2: Pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 2
  Day 2: Pre-dose |  |  |  |  |  |  |  |  |  |  | 3.7300 (6.24287) | -0.1600 (4.11536)
  Day 2: number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 4 | 3 | 5 | 0 | 0
  Day 2 | 2.7750 (1.84369) | 11.2100 (10.32509) | 4.0967 (4.74504) | 8.6233 (11.20869) | 0.1863 (2.04118) | -2.2383 (2.84509) | -0.2317 (0.75466) | 1.7013 (2.56612) | 2.0067 (2.48702) | 2.2360 (4.56081) |  |
  Day 3: Pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2
  Day 3: Pre-dose |  |  |  |  |  |  |  |  |  |  | 2.7583 (7.60588) | -1.8350 (0.65761)
  Day 3: number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 3 | 3.4183 (2.29152) | 11.3767 (5.14516) | 2.3700 (5.72278) | 6.5800 (4.81868) | -1.6687 (3.21471) |  |  |  |  |  |  |
  Day 4: Pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2
  Day 4: Pre-dose |  |  |  |  |  |  |  |  |  |  | 1.8367 (7.00783) | 2.0050 (3.38704)
  Day 5: Pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2
  Day 5: Pre-dose |  |  |  |  |  |  |  |  |  |  | 2.7833 (5.62575) | 0.9100 (4.53963)
  Day 8: Pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 4 | 0 | 0
  Day 8: Pre-dose |  |  |  |  |  | -0.9883 (0.65929) | -0.8617 (2.50250) | 1.9033 (3.87243) | -5.0133 (6.39082) | 4.8563 (3.87653) |  |
  Day 8: 6 hours post-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 4 | 0 | 0
  Day 8: 6 hours post-dose |  |  |  |  |  | -3.0250 (2.66540) | 0.7650 (4.12427) | 2.6400 (3.60712) | -5.2500 (13.55809) | 1.7488 (4.61824) |  |
  Day 8: number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 8 | -1.2350 (3.02842) | 9.1867 (1.78340) | 0.8533 (0.96144) | 2.2867 (3.15587) | -0.9512 (3.31965) |  |  |  |  |  |  |
  Day 9: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 4 | 0 | 0
  Day 9 |  |  |  |  |  | -0.2550 (3.32058) | -1.9250 (1.44439) | 0.9800 (2.77307) | -0.3067 (3.83939) | 2.4963 (3.58692) |  |
  Day 11: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2
  Day 11 |  |  |  |  |  |  |  |  |  |  | 1.0567 (2.53699) | -0.8450 (3.14663)
  Day 15: Pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 4 | 0 | 0
  Day 15: Pre-dose |  |  |  |  |  | 1.4783 (4.88812) | -2.2750 (3.35929) | 3.2767 (2.85037) | -7.0867 (3.29160) | 0.2438 (4.78050) |  |
  Day 15: 6 hours post-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 4 | 0 | 0
  Day 15: 6 hours post-dose |  |  |  |  |  | -1.9083 (4.30519) | -0.8350 (0.48210) | 3.5100 (2.36540) | -3.0233 (10.09021) | 3.6763 (2.82176) |  |
  Day 15: number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 15 | -0.2383 (3.63470) | 5.5633 (1.21378) | -2.3233 (1.80292) | 0.4833 (5.25663) | 0.5763 (1.57608) |  |  |  |  |  |  |
  Day 16: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 4 | 0 | 0
  Day 16 |  |  |  |  |  | -2.6017 (3.59609) | -4.4217 (0.24322) | 1.6800 (1.39796) | -3.9033 (6.24793) | 2.5388 (5.43594) |  |
  Day 18: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2
  Day 18 |  |  |  |  |  |  |  |  |  |  | 0.1600 (1.78332) | -1.3700 (0.77782)
  Day 22: Pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 4 | 0 | 0
  Day 22: Pre-dose |  |  |  |  |  | -3.4417 (0.79907) | -2.5317 (3.12407) | 1.0433 (2.61190) | -3.5567 (3.44181) | 1.6863 (6.44122) |  |
  Day 22: 6 hours post-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 4 | 0 | 0
  Day 22: 6 hours post-dose |  |  |  |  |  | -4.4150 (1.30844) | -3.1183 (2.60335) | 1.4033 (2.70263) | -3.2933 (8.33613) | 4.9788 (8.56683) |  |
  Day 23: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 4 | 0 | 0
  Day 23 |  |  |  |  |  | -2.5650 (2.27414) | -3.5550 (1.42163) | 2.6233 (5.05601) | -3.1900 (6.42324) | 0.7463 (8.20475) |  |
  Day 29: Pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 3 | 3 | 4 | 0 | 0
  Day 29: Pre-dose |  |  |  |  |  | -4.1350 (1.25896) | -2.9725 (3.42593) | 0.1667 (1.82582) | -5.7133 (2.39036) | 2.9863 (9.33491) |  |
  Day 29: 6 hours post-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 3 | 3 | 4 | 0 | 0
  Day 29: 6 hours post-dose |  |  |  |  |  | -4.7350 (0.70326) | 0.3125 (0.06010) | 0.8467 (1.79528) | 0.0567 (11.03200) | 2.7563 (4.51659) |  |
  Day 29: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 29 | 3.0983 (4.90188) | 4.6633 (4.65445) | 2.5133 (5.06806) | -5.2633 (13.06648) | 0.7517 (4.27498) |  |  |  |  |  |  |
  Day 30: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 3 | 3 | 4 | 0 | 0
  Day 30 |  |  |  |  |  | -3.2717 (4.61490) | -4.7375 (3.98455) | 4.8000 (5.94778) | 1.1667 (8.98756) | 0.9888 (7.33033) |  |
  Day 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2
  Day 32 |  |  |  |  |  |  |  |  |  |  | 4.8550 (6.05264) | -0.1150 (4.49013)
  Day 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 3 | 3 | 4 | 0 | 0
  Day 36 |  |  |  |  |  | -0.9383 (2.30022) | -2.2975 (2.85318) | -0.7733 (5.20926) | -3.5333 (8.93039) | 4.8463 (8.26378) |  |
  Day 43: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 3 | 3 | 4 | 0 | 0
  Day 43 |  |  |  |  |  | -3.2550 (0.69262) | -0.0050 | -2.0367 (6.75614) | -3.1533 (3.50810) | 5.1363 (7.51406) |  |
  Day 57: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 3 | 3 | 4 | 0 | 0
  Day 57 |  |  |  |  |  | -5.5517 (4.38918) | 1.0750 | 1.9500 (1.02103) | -7.1667 (9.31929) | 0.4288 (5.91134) |  |

ADVERSE EVENTS:
Time Frame: Serious adverse events (AEs), other AEs and all-cause mortality (deaths) were collected from the first dose of study treatment administration (Day 1) up to 48 weeks (end of the follow-up period) after the last dose of study treatment administration (Part A: Day 337, Part B: Day 365 and Part D: Day 341)
Description: Analysis was performed on the safety analysis set.
Groups:
- Part A - SAD Group1: MRT5005 8 mg: Participants received single dose of MRT5005 8 mg by nebulization on Day1.
- Part A - SAD Group 2: MRT5005 16 mg: Participants received single dose of MRT5005 16 mg by nebulization on Day1.
- Part A - SAD Group 3: MRT5005 20 mg: Participants received single dose of MRT5005 20 mg by nebulization on Day1.
- Part A - SAD Group 4: MRT5005 24 mg: Participants received single dose of MRT5005 24 mg by nebulization on Day1.
- Part B - MAD Group 1: MRT5005 8 mg: Participants received MRT5005 8 mg once weekly by nebulization for 5weeks (i.e., on Day1, Day 8, Day 15, Day 22 and Day 29).
- Part B - MAD Group 3: MRT5005 20 mg: Participants received MRT5005 20 mg once weekly by nebulization for 5 weeks (i.e., on Day 1, Day 8, Day 15, Day 22 and Day 29).
Arm/Group | Part A - SAD Group1: MRT5005 8 mg | Part A - SAD Group 2: MRT5005 16 mg | Part A - SAD Group 3: MRT5005 20 mg | Part A - SAD Group 4: MRT5005 24 mg | Part A - SAD Groups: Pooled Placebo | Part B - MAD Group 1: MRT5005 8 mg | Part B - MAD Group 2: MRT5005 12 mg | Part B - MAD Group 3: MRT5005 16 mg | Part B - MAD Group 3: MRT5005 20 mg | Part B - MAD Groups: Pooled Placebo | Part D: MRT5005 4 mg | Part D: Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/4 | 0/3 | 0/3 | 0/4 | 0/3 | 0/5 | 0/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 1/3 | 1/3 | 3/4 | 1/3 | 1/3 | 0/4 | 2/3 | 2/5 | 1/6 | 1/2
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 4/4 | 3/3 | 3/3 | 4/4 | 3/3 | 5/5 | 6/6 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A - SAD Group1: MRT5005 8 mg (N=3) | Part A - SAD Group 2: MRT5005 16 mg (N=3) | Part A - SAD Group 3: MRT5005 20 mg (N=3) | Part A - SAD Group 4: MRT5005 24 mg (N=3) | Part A - SAD Groups: Pooled Placebo (N=4) | Part B - MAD Group 1: MRT5005 8 mg (N=3) | Part B - MAD Group 2: MRT5005 12 mg (N=3) | Part B - MAD Group 3: MRT5005 16 mg (N=4) | Part B - MAD Group 3: MRT5005 20 mg (N=3) | Part B - MAD Groups: Pooled Placebo (N=5) | Part D: MRT5005 4 mg (N=6) | Part D: Placebo (N=2)
Infective Pulmonary Exacerbation Of Cystic Fibrosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (4) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 1 (3) | 1 (2)
Anaphylactic Reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis Acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus Urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A - SAD Group1: MRT5005 8 mg (N=3) | Part A - SAD Group 2: MRT5005 16 mg (N=3) | Part A - SAD Group 3: MRT5005 20 mg (N=3) | Part A - SAD Group 4: MRT5005 24 mg (N=3) | Part A - SAD Groups: Pooled Placebo (N=4) | Part B - MAD Group 1: MRT5005 8 mg (N=3) | Part B - MAD Group 2: MRT5005 12 mg (N=3) | Part B - MAD Group 3: MRT5005 16 mg (N=4) | Part B - MAD Group 3: MRT5005 20 mg (N=3) | Part B - MAD Groups: Pooled Placebo (N=5) | Part D: MRT5005 4 mg (N=6) | Part D: Placebo (N=2)
Acute Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Candida Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infective Pulmonary Exacerbation Of Cystic Fibrosis (Infections and infestations) | 3 (4) | 2 (2) | 3 (4) | 3 (8) | 3 (10) | 3 (8) | 0 (0) | 2 (4) | 0 (0) | 2 (3) | 3 (6) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mycobacterial Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis Media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis Streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinovirus Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sialoadenitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (2)
Systemic Candida (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral Rash (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal Mycotic Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Allergy To Vaccine (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Increased Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Attention Deficit Hyperactivity Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anosmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disturbance In Attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 3 (4) | 1 (1) | 3 (6) | 1 (1) | 1 (1) | 1 (3) | 1 (4) | 3 (10) | 1 (1) | 2 (3) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental Impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy Peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep Paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye Pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision Blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperaemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (11) | 2 (4) | 1 (1) | 3 (7) | 0 (0) | 3 (12) | 2 (2) | 4 (8) | 1 (2) | 3 (7) | 2 (2) | 2 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 2 (3) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Increased Bronchial Secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased Upper Airway Secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Paranasal Sinus Discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paranasal Sinus Hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiration Abnormal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus Polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sputum Discoloured (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sputum Increased (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (6) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain Lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dental Caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epigastric Discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric Polyps (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal Motility Disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingival Swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertrophy Of Tongue Papillae (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth Deposit (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ingrowing Nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail Pigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night Sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (4) | 0 (0)
Trigger Finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glycosuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Morning Sickness (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast Pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspareunia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine Pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal Discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Discomfort (General disorders) | 1 (3) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (4) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 2 (6) | 0 (0) | 1 (1) | 0 (0)
Crepitations (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Feeling Abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection Site Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 2 (6) | 0 (0) | 0 (0) | 0 (0)
Reactogenicity Event (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaccination Site Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Creatinine Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Uric Acid Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body Temperature Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breath Sounds Abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
C-Reactive Protein Increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Forced Expiratory Volume Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungal Test Positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart Rate Irregular (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic Enzyme Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes Simplex Test Positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver Function Test Abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mycobacterium Test Positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pulmonary Function Test Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sputum Abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Streptococcus Test Positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Burns First Degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament Sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2020-07-30): https://cdn.clinicaltrials.gov/large-docs/47/NCT03375047/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/47/NCT03375047/SAP_001.pdf